CLINICAL TRIAL: NCT07357480
Title: Comparison of Target-Controlled Infusion Using the Eleveld Model and Manual Total Intravenous Anesthesia on Intraoperative Anesthetic Consumption and Postoperative Pain and Delirium in Supratentorial Surgery
Brief Title: Comparison of Target-Controlled and Manual Total Intravenous Anesthesia in Supratentorial Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ali Okuyan, Research Assistant, Department of Anesthesiology and Reanimation, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-24687260-604.01-1504004
Record Dates: First submitted 2026-01-10; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Delirium (POD); Postoperative Pain; PONV; Burst Suppression; Recovery Period, Anesthesia
Keywords: Target Controlled Infusion; Total Intravenous Anesthesia; Eleveld Model; Postoperative Delirium; Supratentorial Surgery; Bispectral Index; Propofol; Remifentanil
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups to receive either target-controlled infusion or manually controlled total intravenous anesthesia.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Total Intravenous Anesthesia (Experimental): Participants receive manually controlled total intravenous anesthesia using propofol and remifentanil, with dosing adjusted by the anesthesiologist based on clinical parameters and bispectral index monitoring.
  Interventions: Device: Total Intravenous Anesthesia(TIVA)
- Target-Controlled Infusion (TCI) (Experimental): Participants receive target-controlled infusion of propofol and remifentanil using the Eleveld pharmacokinetic model, with effect-site targeting throughout the surgical procedure.
  Interventions: Device: Target Controlled Infusion

INTERVENTIONS:
Device: Target Controlled Infusion — Total Intravenous Anesthesia (TIVA) will be administered using an infusion pump (e.g., BeneFusion nSP) equipped with the Eleveld pharmacokinetic model. Propofol will be initiated at a target concentration of 3-3.5 µg/ml, and Remifentanil at 2-3 ng/ml (effect-site targeting). The "opioid present" option will be selected for the propofol model. Doses will be titrated to maintain a Bispectral Index (BIS) value between 40-60 throughout the surgery.
  Arms: Target-Controlled Infusion (TCI)
Device: Total Intravenous Anesthesia(TIVA) — Total Intravenous Anesthesia (TIVA) will be administered via manual titration. Induction will be performed with 20 mg propofol boluses based on EEG changes on the BIS monitor, followed by a remifentanil infusion of 0.1 µg/kg/min. Maintenance doses will be manually adjusted by the anesthesiologist to maintain a Bispectral Index (BIS) value between 40-60 and hemodynamic stability.
  Other Names: Manually controlled Total Intravenous Anesthesia
  Arms: Manual Total Intravenous Anesthesia

SUMMARY:
This study aims to investigate the effect of target-controlled infusion using the Eleveld pharmacokinetic model compared with manually controlled total intravenous anesthesia on the incidence of postoperative delirium in patients undergoing supratentorial surgery. Propofol and remifentanil are administered using either target-controlled or manual infusion techniques according to the study protocol. Secondary objectives include comparisons of intraoperative anesthetic consumption, hemodynamic responses, recovery profiles, postoperative pain, and postoperative nausea and vomiting between the two anesthesia strategies. The study seeks to evaluate whether target-controlled infusion provides improved anesthetic management and postoperative outcomes compared with manual total intravenous anesthesia.

DETAILED DESCRIPTION:
This study will be conducted following approval by the Istanbul University-Cerrahpaşa Medical Research Ethics Committee (Approval No: 1504004) in patients scheduled for supratentorial craniotomy at the operating rooms of the Department of Neurosurgery, Cerrahpaşa Faculty of Medicine, Istanbul University-Cerrahpaşa, after obtaining written informed consent. The study is designed as a prospective, randomized controlled trial with two groups: a manually controlled total intravenous anesthesia group (Manual group) and a target-controlled infusion group (TCI group).

Sample size calculation was performed based on the delirium rates reported in the study by Varsha, as no direct comparison between target-controlled infusion and manual total intravenous anesthesia in terms of delirium was identified in the available literature. In that study, the incidence of postoperative delirium was reported as 34.2% (12/35) in the inhalational anesthesia group and 8.8% (3/34) in the propofol total intravenous anesthesia group. Based on these proportions, an a priori power analysis was conducted using G*Power version 3.1.9.7 for comparison of proportions between two independent groups. Assuming a one-sided test, an alpha level of 0.05, power of 80% (1-β = 0.80), and a group allocation ratio of N2/N1 = 0.97, a minimum of 32 patients in the first group and 31 patients in the second group were required, resulting in a total sample size of 63 patients.

Adult male and female patients aged 18-60 years undergoing supratentorial surgery and classified as American Society of Anesthesiologists (ASA) physical status I or II will be included. Exclusion criteria include refusal to provide consent, ASA physical status III or higher, pregnancy, emergency surgery, presence of brain herniation, anticipated or documented difficult airway, inability to communicate (non-Turkish speaking or hearing impairment), preoperative risk factors for delirium (substance abuse, use of neuropsychiatric medications, preoperative hemoglobin concentration below 8 g/dL, malnutrition, electrolyte or thyroid hormone abnormalities), intraoperative deviations from the study protocol (changes in surgical or anesthetic technique, severe intraoperative complications), and contraindications to propofol or remifentanil use.

Eligible patients will be randomized into either the Manual Total Intravenous Anesthesia group or the Target-Controlled Infusion group using the sealed-envelope method. Patient evaluation will begin during routine preoperative anesthesia assessment, including screening for delirium using the Confusion Assessment Method (CAM). In the operating room, in addition to standard monitoring, bispectral index monitoring (BIS™, Covidien/Medtronic, USA), invasive arterial blood pressure monitoring, and bladder catheterization will be applied to all patients. Demographic data and baseline hemodynamic measurements (blood pressure and heart rate) will be recorded prior to induction of anesthesia.

Anesthesia induction will be performed using remifentanil, propofol, and rocuronium. To reduce injection pain associated with propofol, 40 mg intravenous lidocaine will be administered using a tourniquet technique. In the Manual group, after initiation of remifentanil infusion at 0.1 µg/kg/min, propofol will be administered in 20-mg boluses guided by electroencephalographic changes observed on the BIS monitor. In the TCI group, automatic induction will be performed using an infusion pump (BeneFusion nSP, Mindray Bio-Medical Electronics Co., China) with target concentrations of 2-3 ng/mL for remifentanil and 3-3.5 µg/mL for propofol. For both drugs, the Eleveld pharmacokinetic model with effect-site targeting will be used, and opioid co-infusion mode will be enabled for propofol administration. In both groups, rocuronium at a dose of 0.6-0.9 mg/kg will be administered intravenously once delta waves are observed on the raw EEG display of the BIS monitor, followed by tracheal intubation.

During the induction period, induction time, total propofol dose, immediate post-intubation monitoring data, and burst suppression duration will be recorded. Induction time will be defined as the interval between initiation of propofol administration and the appearance of delta waves on the BIS monitor. Following intubation, scalp block using 15-20 mL of 0.5% bupivacaine, intravenous dexketoprofen 50 mg, and antibiotic prophylaxis will be administered when not contraindicated. Mechanical ventilation will be provided using a volume-controlled mode with AutoFlow enabled (VC-AF) via an anesthesia workstation (Perseus A500, Dräger, Lübeck, Germany), with tidal volumes of 4-8 mL/kg and positive end-expiratory pressure of 5-8 cmH₂O.

Anesthesia maintenance in both groups will be achieved using propofol-remifentanil total intravenous anesthesia. In patients not undergoing intraoperative neuromonitoring, rocuronium infusion at 20-30 mg/h will be administered. Propofol and remifentanil doses will be titrated by the attending anesthesiologist to maintain BIS values between 40 and 60 and to achieve normotension. Total propofol and remifentanil consumption and burst suppression durations will be recorded at the 1st, 2nd, and 4th intraoperative hours and at the end of surgery. At the conclusion of surgery, patients will receive intravenous tramadol (50-100 mg), ondansetron (8 mg), and sugammadex (200 mg). Patients who are not clinically suitable for extubation will be transferred to the intensive care unit intubated and excluded from the study.

During the extubation period, time to awakening, extubation time, post-extubation monitoring data, total drug consumption, total burst suppression duration, and surgical and anesthesia durations will be recorded. Awakening time will be defined as the interval between discontinuation of infusions and the patient's response to verbal commands, and extubation time as the interval between infusion cessation and tracheal extubation.

The recovery period will be defined as the first postoperative hour. Hemodynamic measurements, pain intensity assessed using the Numeric Rating Scale (NRS), presence of nausea and vomiting, recovery profile assessed using the Aldrete score, and additional analgesic requirements will be recorded at 15, 30, and 60 minutes postoperatively. Patients in both groups will be followed for postoperative delirium for three days. Delirium assessments will be performed using CAM at postoperative hour 6, at 08:00 on the first postoperative day, and at 24, 48, and 72 hours postoperatively. For patients discharged before 72 hours, the final assessment will be conducted at discharge.

Due to the nature of the study, the attending anesthesiologist will be aware of group allocation during the intraoperative period. However, postoperative recovery and delirium assessments will be performed by a nurse and/or physician blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 60 years
* Scheduled for elective supratentorial surgery under general anesthesia
* American Society of Anesthesiologists (ASA) physical status I or II
* Planned total intravenous anesthesia with propofol and remifentanil
* Ability to provide written informed consent

Exclusion Criteria:

* Refusal or inability to provide written informed consent
* American Society of Anesthesiologists (ASA) physical status III or higher
* Pregnancy
* Emergency surgery
* Presence of brain herniation
* Anticipated or documented difficult airway
* Inability to communicate effectively (e.g., non-Turkish speaking or hearing impairment)
* Preoperative risk factors for delirium, including substance abuse, use of neuropsychiatric medications, preoperative hemoglobin level < 8 g/dL, malnutrition, or electrolyte or thyroid hormone abnormalities
* Intraoperative deviation from the study protocol, including changes in surgical or anesthetic technique or occurrence of major intraoperative complications
* Contraindications to propofol or remifentanil

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Delirium | Postoperative 72 hours
  Postoperative delirium will be assessed using the Confusion Assessment Method (CAM) during the first 72 hours after surgery

SECONDARY OUTCOMES:
Total Propofol and Remifentanil Consumption | Intraoperative period
  The total amount of propofol and remifentanil administered intraoperatively will be recorded and compared between the study groups
Heart rate | Intraoperative period
  Heart rate will be recorded as beats per minute intraoperatively and compared between groups
Blood pressure | Intraoperatively
  Blood pressure will be recorded as mmHg intraoperatively and compared between groups
Burst Suppression Duration | Intraoperative period
  The total duration of burst suppression observed on bispectral index monitoring during anesthesia will be recorded
Recovery Profile | From discontinuation of anesthetic infusion until 1 hour after extubation
  Recovery characteristics, including time to awakening and time to extubation, will be assessed and compared between groups
Postoperative Pain | First postoperative hour
  Postoperative pain severity will be assessed using the Numeric Rating Scale (NRS) between 0-10, (higher means more pain)
Postoperative Nausea and Vomiting | First postoperative hour
  The presence of postoperative nausea and vomiting will be recorded during the early postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Ali Okuyan, MD, Principal Investigator — İstanbul University-Cerrahpaşa, Cerrahpaşa Medical Faculty
Locations (1):
- Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this is a single-center academic thesis study and data sharing was not included in the informed consent

REFERENCES:
- [Background] Daccache N, Wu Y, Jeffries SD, Zako J, Harutyunyan R, Pelletier ED, Laferriere-Langlois P, Hemmerling TM. Safety and recovery profile of patients after inhalational anaesthesia versus target-controlled or manual total intravenous anaesthesia: a systematic review and meta-analysis of randomised controlled trials. Br J Anaesth. 2025 May;134(5):1474-1485. doi: 10.1016/j.bja.2025.02.007. Epub 2025 Mar 11. PMID 40074622
- [Background] Varsha AV, Unnikrishnan KP, Saravana Babu MS, Raman SP, Koshy T. Comparison of Propofol-Based Total Intravenous Anesthesia versus Volatile Anesthesia with Sevoflurane for Postoperative Delirium in Adult Coronary Artery Bypass Grafting Surgery: A Prospective Randomized Single-Blinded Study. J Cardiothorac Vasc Anesth. 2024 Sep;38(9):1932-1940. doi: 10.1053/j.jvca.2024.05.027. Epub 2024 May 23. PMID 38987101